CLINICAL TRIAL: NCT03124524
Title: Which do You Think is the Best Treatment Choice in Primary Dysmenorrhea?
Brief Title: Treatment Choice in Primary Dysmenorrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Adana Numune Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gulsum Uysal, Principal Investigator, MD., Adana Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/290
Record Dates: First submitted 2017-03-09; First posted 2017-04-24 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Primary Dysmenorrhea
Keywords: estradiol valerate/dienogest; ethinylestradiol/ drospirenone; pelvic pain; primary dysmenorrhea; uterine artery doppler indices
MeSH Terms: conditions — Pelvic Pain | interventions — estradiol valerate-dienogest; Ethinyl Estradiol; drospirenone; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): 33 healthy controls
- Qlarista Group (Active Comparator): group who were administered estradiol valerate/dienogest
  Interventions: Drug: estradiol valerate/dienogest
- Yasmin Group (Active Comparator): group who were administered ethinylestradiol and drospirenone
  Interventions: Drug: ethinylestradiol and drospirenone

INTERVENTIONS:
Drug: estradiol valerate/dienogest — oral, 28 tablets including 2 tablets of 3mg estradiol valerate, 5 tablets of 2mg estradiol valerate plus 2mg dienogest, 17 tablets of 2mg estradiol valerate plus 3mg dienogest, 2 tablets of 1mg estradiol valerate and 2 non hormonal tablets as placebo, respectively
  Other Names: Qlarista; Bayer HealthCare Berlin, Germany
  Arms: Qlarista Group
Drug: ethinylestradiol and drospirenone — oral,0.03 mg ethinylestradiol and 3 mg drospirenone (21 tablets)
  Other Names: Yasmin; Bayer HealthCare Berlin, Germany
  Arms: Yasmin Group

SUMMARY:
Our aim is to evaluate and compare the pain relief of estradiol valerate/dienogest and ethinylestradiol/ drospirenone by using doppler indices.

100 nullipara patients with symptoms of severe primary dysmenorrhea (PD) requesting contraception aged from 18 to 35 were included to the study. Visual analog scale (VAS), the uterine artery doppler indices including systole/diastole rates ( S/D), pulsatility index (PI) and resistance index (RI) values were evaluated and recorded in both uterine vessels before treatment. The 66 PD patients who met the inclusion criteria were divided into 2 groups and 33 healthy controls created Group 1. Group 2 were administered estradiol valerate/dienogest while Group 3 were administered 0.03 mg ethinylestradiol and 3 mg drospirenone. Both VAS scores and doppler indices were repeated after 3 months treatment. The changes in values were recorded.

DETAILED DESCRIPTION:
This prospective, randomized, controlled clinical trial was conducted in Kayseri Education and Research Hospital, in Turkey between 2015 and 2016. Nullipara patients with symptoms of severe primary dysmenorrhea (PD) requesting contraception aged from 18 to 35 were included to the study. Afterwards, based on computer generated random numbers the patients were allocated to one of the two study arms; Group2 (Qlarista group) and Group3 (yasmin group), equally.

The PD was diagnosed clinically. The characteristic of pain was periodic (at least following 3 menstrual cycles), midline, lower abdominal cramps or pelvic colic like pain that starts up to one day before menses, lasts for the 3 days of bleeding, gradually diminishes over 12 to 72 hours and ends after period. The pain starts generally in 2 to 3 years after menarche with regular menses (25-31 day). Also absence of pelvic pathology was important in these patients for diagnosis.

Patients with history of pelvic inflammatory diseases, endometriosis, ovarian cysts, chronic abdominal pain, fibroids, obstructive endometrial polyps, cervical stenosis, inflammatory bowel syndrome, irritable bowel syndrome, major abdominal or pelvic surgery, intrauterine device and congenital obstructive müllerian malformations were excluded. Smoking, overweighted (body mass index (BMI) ≥ 30) patients that oral contraceptive pills (OCP) treatment was contraindicated were also excluded. Additionally, patients enrolled simultaneously into other studies that require drug intake or otherwise prevent compliance with protocol were out of the study.

Visual analog scale (VAS) from 0 (no pain) to 10 (maximum pain, 'worst pain I have ever felt') was applied to patients on the first day of menstrual cycle. Patients with VAS score of between 7 to10 and PD accompanied with vomiting, nausea, dizziness, headache, nervousness, diarrhea and fatigue were classified as severe PD. The ages (years), BMI (kg/m2), length of menstrual cycle (days) and length of bleeding (days) and demographic data of patients were recorded.

Before treatment during menstruation period all ultrasound examinations were carried out trans abdominally with Toshiba Xario machine ( Shimoishigami, Otawara-shi, Tochigi 324-8550, Japan) equipped with a 2.8-7 megahertz (MHz) transducer by a single radiologist (Ş.T.) The uterine artery blood flows were measured at the lateral level of uterine artery neighbour to cervicocorporeal junction in both sides (right and left). Doppler indices including systole/diastole rates ( S/D), pulsatility index (PI) and resistance index (RI) values were evaluated and recorded in both uterine vessels. Both VAS scores and doppler indices were repeated after 3 months treatment. The changes in values were recorded.

According to previously published studies and after power analyses, when α error and β error were considered, respectively, as 0.05 and 0.20, with 80% power number of patients for each group were determined as minimum 30. Power Analysis and Sample Size Software (PASS) 11 software (NCSS, Kaysville, USA) was used to perform these analyses. Regarding dropout rates (40 % -50 %) in similar studies over the treatment period we planned to include 100 patients with PD and 40 healthy controls. The PD patients who met the inclusion criteria were divided into 2 groups. Patients in Group 2 were administered estradiol valerate/dienogest (Qlarista; Bayer HealthCare Berlin, Germany). Qlarista consists of 28 tablets (including 2 tablets of 3mg estradiol valerate, 5 tablets of 2mg estradiol valerate plus 2mg dienogest, 17 tablets of 2mg estradiol valerate plus 3mg dienogest, 2 tablets of 1mg estradiol valerate and 2 non hormonal tablets as placebo, respectively). Patients in Group 3 were administered 0.03 mg ethinylestradiol and 3 mg drospirenone (21 tablets) (Yasmin; Bayer HealthCare Berlin, Germany). Patients were randomly administered to the 2 treatments in a 1:1 ratio. Instead of relieving, patients were not allowed to use rescue medication (NSAI drugs) to prevent menstruation related pelvic pain.

All procedures performed in studies involving human participants were in accordance with the ethical standards of the institutional and/or national research committee and with the 1964 Helsinki declaration and its later amendments or comparable ethical standards. Ethics approval for the study was obtained from Erciyes University Hospital (protocol number:2014/290). Informed consent was obtained from all patients who included in our study.

All analyses were performed using the SPSS for Windows 21.0 (SPSS Inc. USA) software package. The normality of distribution for variables was assessed using the Shapiro Wilk test. Data was presented as means ± standart deviation (SD) for continuous variables. To assess the differences in variables between groups, the independent t test was used. As the results did not have a normal distribution, Kruskal-Wallis, Mann-Whitney U-test and Bonferroni correction was used in the comparisons between the groups. For comparison, the Wilcoxon test was applied to the results (VAS scores, Doppler flow parameters) before and after receiving therapy. For all comparisons, the P < 0.05 value was determined as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* must be nullipara patients with symptoms of severe primary dysmenorrhea.
* The characteristic of pain must be periodic (at least following 3 menstrual cycles),
* midline,
* lower abdominal cramps or pelvic colic like pain that starts up to one day before menses,
* lasts for the 3 days of bleeding,
* gradually diminishes over 12 to 72 hours,
* ends after period.
* The pain must start generally in 2 to 3 years after menarche with regular menses (25-31 day).

Exclusion Criteria:

* Patients with history of pelvic inflammatory diseases,
* endometriosis,
* ovarian cysts,
* chronic abdominal pain,
* fibroids,
* obstructive endometrial polyps,
* cervical stenosis,
* inflammatory bowel syndrome,
* irritable bowel syndrome,
* major abdominal or pelvic surgery,
* intrauterine device,
* congenital obstructive müllerian malformations.
* patients that OCP treatment was contraindicated
* patients enrolled simultaneously into other studies that require drug intake or otherwise prevent compliance with protocol.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2016-10-10 (Actual)

PRIMARY OUTCOMES:
Doppler indices of uterine artery blood flows. | up to 10 minutes
  Before and treatment during menstruation period the uterine artery blood flows were measured at the lateral level of uterine artery neighbour to cervicocorporeal junction in both sides (right and left). Doppler indices including systole/diastole rates ( S/D), pulsatility index (PI) and resistance index (RI) values were evaluated and recorded in both uterine vessels.

SECONDARY OUTCOMES:
Questionnaire Questionarie: Pain relief by using Visual analog scale (VAS) before and after treatment. | up to 10 minutes
  VAS from 0 (no pain) to 10 (maximum pain, 'worst pain I have ever felt') was applied to patients on the first day of menstrual cycle. Patients with VAS score of between 7 to10 and PD accompanied with vomiting, nausea, dizziness, headache, nervousness, diarrhea and fatigue were classified as severe PD. The ages (years), BMI (kg/m2), length of menstrual cycle (days) and lenght of bleeding (days) and demographic data of patients were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gulsum Uysal, M.D, Principal Investigator — Adana Numune Training and Research Hospital

IPD SHARING:
Plan to Share IPD: Yes
if needed